CLINICAL TRIAL: NCT02774148
Title: Pain Control in Elderly Hip Fracture Patients: Is Intravenous Acetaminophen Superior to Oral Administration?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Proved difficult to consent patient population due to comorbidities
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-225
Record Dates: First submitted 2016-05-09; First posted 2016-05-17 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PO Acetaminophen (Active Comparator): 1,000mg Acetaminophen po every 8 hours until discharge.
  Interventions: Drug: PO Acetaminophen
- IV Acetaminophen (Experimental): 1,000mg Acetaminophen IV every 8 hours until the patient has received 3 doses post-operatively. Then 1,000mg Acetaminophen po every 8 hours until discharge.
  Interventions: Drug: IV Acetaminophen

INTERVENTIONS:
Drug: IV Acetaminophen — The patient will receive 1,00mg IV Acetaminophen every 8 hours until 3 doses have been received post-operatively.
  Other Names: Ofirmev
  Arms: IV Acetaminophen
Drug: PO Acetaminophen — The patient will receive 1,000mg po Acetaminophen every 8 hours.
  Other Names: Tylenol
  Arms: PO Acetaminophen

SUMMARY:
The primary objective is to determine if intravenous acetaminophen decreases pain scores and the amount of morphine equivalence received as compared to oral acetaminophen in patients greater than 65 years old after sustaining a hip fracture.

DETAILED DESCRIPTION:
Surgeons involved in this research agree to the randomization of patients into one of two groups. After informed consent, patients will be randomly assigned in a 1:1 ratio to the treatment group or the control group.

Group 1: This group will serve as the control group, and will be scheduled to receive one gram (1g) acetaminophen PO every 8 hours.

Group 2: This group will serve as the treatment group, and will be scheduled to receive one gram (1g) acetaminophen IV every 8 hours

The standardized pain control protocol for hip fracture patients will be initiated for all patients. The pain protocol will be initiated at hospital admission, and after three postoperative doses of the group assigned acetaminophen all patients will be switched to one gram scheduled acetaminophen PO in preparation for hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Acute, isolated, unilateral femoral neck, intertrochanteric, and per trochanteric hip fractures confirmed by anteroposterior/lateral hip radiographs, computed tomography, or magnetic resonance imaging (MRI).
2. Age ≥ 65 years.
3. Low energy mechanism.
4. Hip fracture fixation performed within 48 hours of injury.
5. English speaking.
6. Anticipated medical optimization for operative fixation.
7. No other major trauma.

Exclusion Criteria:

1. Unable to provide informed consent (dementia, limited decision making capacity)
2. Admitted by medical service for significant co-morbidities
3. Retained hardware around the affected hip
4. Infection around the affected hip
5. Transfer patients with a length of stay > 24 hours at the transferring hospital
6. Known allergy to acetaminophen
7. Current use of narcotics
8. Receiving a regional anesthetic block at any point during the hospitalization
9. Known history of hepatic disease (hepatitis, cirrhosis)
10. Weight < 50kg
11. Prisoner
12. Involved in another clinical trial that would interfere with the intervention of this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R. Fras, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PO Acetaminophen | IV Acetaminophen
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one patient was enrolled, therefore data was not sufficient to run an analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | PO Acetaminophen | IV Acetaminophen | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Pain scores will be compared between the two groups.
Time Frame: 6 days
Population: No analyses complete due to early termination.
Arm/Group | PO Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Amount of Morphine Equivalents, as Determined by an Opioid Dose Calculator, Received by the Patient.
Description: The amount of opioid pain medication a patient receives will be recorded and the Morphine equivalents will be determined by an opioid dose calculator. The morphine equivalents will be compared between the two groups.
Time Frame: 6 days
Population: No analyses complete due to early termination.
Arm/Group | PO Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Timing of First Day of Ambulation.
Description: The timing of the first day of ambulation will be compared between the two groups.
Time Frame: 6 days
Population: No analyses complete due to early termination.
Arm/Group | PO Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Distance Ambulated
Description: The distance ambulated will be compared between the two groups.
Time Frame: 6 days
Population: No analyses complete due to early termination.
Arm/Group | PO Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Hospital Stay
Description: Length of hospital stay will be compared between the two groups.
Time Frame: 2 weeks
Population: No analyses complete due to early termination.
Arm/Group | PO Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | PO Acetaminophen | IV Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to difficulty enrolling patient population and limitations due to timing required to consent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes